CLINICAL TRIAL: NCT01324414
Title: Predictive Value of Inflammation and Fibrosis in Skeletal Muscle for Liver Histopathology in Patients With Non Alcoholic Fatty Liver Disease: Impact of Muscle Insulin Resistance on the Pathogenesis of Non Alcoholic Steatohepatitis
Brief Title: Impact of Muscle Insulin Resistance on the Pathogenesis of Non Alcoholic Steatohepatitis
Acronym: NASHCR20
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bashar Aqel, MD, Mayo Clinic
Other Study IDs: 10-002215
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Non Alcoholic Fatty Liver Diseases (NAFLD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of Non alcoholic fatty liver disease (NAFLD) continues to increase, and prevalence estimates for NAFLD range from 17-33%, making it is the most common cause of chronic liver disease in North America. It is associated with increased cardiovascular morbidity as well as progression to cirrhosis is a subset of patients. There is currently no approved treatment for NAFLD. A key barrier to the development of effective therapies is a lack of consensus on the criteria for diagnosis and endpoints for studies evaluating diagnostic markers, prognosis and therapeutic modalities.

NAFLD encompasses an entire pathological spectrum of disease, from relatively benign accumulation of lipid (steatosis) to progressive non alcoholic steatohepatitis (NASH) associated with inflammation, fibrosis, and necrosis. It has been estimated that 20-30% of patients with NAFLD will exhibit biochemical and histological changes characteristic of NASH, and 15-20% of those patients will progress to have cirrhosis. NASH remains an important phenotypic state, because this sub-group of patients is deemed at high-risk for developing progressive disease resulting in cirrhosis, liver failure requiring transplantation, or death.

Although NAFLD has not to date been included as a component of the metabolic syndrome, there is increasing evidence that NAFLD frequently accompanies the development of insulin resistance and therefore may be an indicator or predictor of future cardiometabolic risk. Moreover, recent findings in skeletal muscle of experimental insulin resistance (lipid infusion) as well as naturally occurring obese and type 2 diabetic, insulin resistant patients show that skeletal muscle inflammation leads to a pattern of extracellular matrix, structural, and remodeling abnormalities that closely resemble the TGFb, connective tissue growth factor (CTGF) mediated fibrotic response that differentiates simple steatotic liver from NASH. This suggests there may be a common underlying mechanism. Given the ready availability of skeletal muscle tissue using percutaneous needle muscle biopsies, compared to the more invasive liver biopsy, it may be possible to use characteristics of skeletal muscle to distinguish the severity of liver fibrosis.

Given the preponderance of patients being identified with NAFLD, the recognition of less and non invasive tests that help to discriminate the different phenotypic types of NAFLD would be highly practical and useful. This would help identify patients at risk of progression to cirrhosis, and thus make them the target of any available therapeutic interventions.

The investigators hypothesize that 1. Insulin resistance measured through glucose tolerance test directly correlates with the extent of liver and muscle fibrosis, and 2. Inflammation and fibrosis in the skeletal muscles correlates with the histopathological changes seen in patients with NAFLD, and potentially skeletal muscle inflammation may be used as a diagnostic predictor to differentiate patients with NASH from patients with simple steatosis.

The overall goal of this project is to determine the extent to which inflammation and fibrosis in skeletal muscle mirrors and is predictive of the level of liver inflammation and can distinguish NASH from simple steatosis. Specifically, the investigators propose the following Aims:

1. To use estimates of insulin sensitivity from modeling of oral glucose tolerance tests to test the hypothesis that the extent of liver and muscle fibrosis is directly related to insulin resistance.
2. To use liver and muscle biopsies to characterize the changes in abundance of mRNAs and proteins that characterize inflammation, extracellular matrix remodeling, and fibrosis. The investigators will use quantitative rt-PCR and immunoblot analysis to compare mRNA expression and protein abundance of collagens I and III, fibronectin, and connective tissue growth factor (CTGF) to test the hypothesis that there is a direct relationship between the levels of these proteins in muscle and liver and the degree of fibrosis.
3. To establish a biospecimen repository of serum, mRNA from circulating white blood cells, liver and muscle tissue, and DNA to serve as the substrate for future studies of the pathogenesis of NASH.

ELIGIBILITY:
Inclusion Criteria:

Ability and willingness to give written, informed consent to be screened for and if eligible to be enrolled in the study.

* Age > 18 years old.
* Minimal or no alcohol use (< 14 drinks/week in a man, < 7 drinks/week in a woman. Approximately 10g of alcohol equals one drink unit. One drink unit equals 1 ounce of distilled spirit, one 12-oz beer, or one 4-oz glass of wine.
* Collection of a standard of care liver biopsy that is obtained within 120 days of enrollment.
* Collection of biosamples (serum, plasma, PMNC, muscle biopsy) within 90 days of enrollment.
* NAFLD diagnosis based on standard clinical, imaging, and histological criteria.

Exclusion Criteria:

* Pregnant women.
* Age < 18 years old.
* Unable to consent for study.
* Patients who underwent liver transplant.
* Patients on oral steroids for more than 2 weeks within 6 months of enrollment.
* Patients with Diabetes Mellitus.
* Clinical or histological evidence of alcoholic liver disease: Regular and excessive alcohol use within two years of enrollment: > 14 drinks/week in a man, >7 drinks/week in a woman.
* Absence of any other liver disease: Autoimmune hepatitis, viral hepatitis, alpha-1 antitrypsin deficiency, hemochromatosis, drug induced liver injury, Wilson's disease, or cholestatic liver disease.
* Known HIV.
* Hepatocellular carcinoma.
* History of bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with NAFLD
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Identification of a unique skeletal muscle histopathology, specific tissue, genomic markers and muscle pathophysiology that help to differentiate patients with NASH from those with simple steatosis | Three months

SECONDARY OUTCOMES:
Determination of insulin resistance and sensitivity in patients with NAFLD who do not have diabetes mellitus | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Bashar Aqel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States